CLINICAL TRIAL: NCT03665987
Title: The Effect of Preoperative Assessment Clinic on Prognosis and Economic Results of Patients With Coexisting Diseases.
Brief Title: The Effect of Preoperative Assessment Clinic on Prognosis and Economic Results of Patients With Coexisting Disease.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2018-112R
Record Dates: First submitted 2018-09-01; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Length of Stay; Postoperative Complications; Morality
MeSH Terms: conditions — Postoperative Complications | interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- properative assessment clinic group: The treatment group will be seen in the preoperative clinic before hospitalization.
  Interventions: Behavioral: consultation in preoperative assessment clinic
- Control group: The control group will get anesthetic consultation after hospitalization without clinic service.

INTERVENTIONS:
Behavioral: consultation in preoperative assessment clinic — The treatment group will be seen in the preoperative clinic before hospitalization, while the control group will get anesthetic consultation after hospitalization without clinic service. No additional interventions will be given during and after surgery.
  Groups: properative assessment clinic group

SUMMARY:
To assess the effect of preoperative assessment clinic on prognosis and economic results of patients with coexisting diseases, the investigators designed a prospective cohort study. The investigators will recruit 250 patients preparing to undergo a selective epigastrium surgery with coexisting medical diseases which need an anesthetic consultation. The patients will be randomly assigned into two groups. The intervention group will be seen in the preoperative clinic before hospitalization, while the control group will get anesthetic consultation after hospitalization without clinic service. No additional interventions will be given during and after surgery. The length of stay, hospitalization expense, postoperative complication rate and mortality rate of the two groups will be compared. The investigator assume that consultation in preoperative assessment clinic will improve the prognosis and decrease the hospitalization expenses.

ELIGIBILITY:
Inclusion Criteria:

* patients preparing to undergo a selective epigastrium surgery
* patients with coexisting medical diseases needing an anesthetic consultation
* over 60 years old
* ASA II-III
* patients with good compliance

Exclusion Criteria:

* patients ubdergoing emergency operation
* ASA I, IV
* patients under 60 years old
* patients with bad compliance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from outpatient surgery department in Shanghai Zhongshan Hospital.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
length of stay | an average of 5 days

SECONDARY OUTCOMES:
hospitalization expense | an average of 5 days
  The expense patients cost during hospitalization

OTHER OUTCOMES:
postoperative complication rate | an average of 5 days
mortality rate | an average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jing Cang, Doctor, Study Chair — Shanghai Zhongshan Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The participants haven't recruited yet and we have no idea about sharing IPD to other reearchers. Maybe we will share the clinical study report to other researchers.

REFERENCES:
- [Result] van Klei WA, Moons KG, Rutten CL, Schuurhuis A, Knape JT, Kalkman CJ, Grobbee DE. The effect of outpatient preoperative evaluation of hospital inpatients on cancellation of surgery and length of hospital stay. Anesth Analg. 2002 Mar;94(3):644-9; table of contents. doi: 10.1097/00000539-200203000-00030. PMID 11867390
- [Result] Ferschl MB, Tung A, Sweitzer B, Huo D, Glick DB. Preoperative clinic visits reduce operating room cancellations and delays. Anesthesiology. 2005 Oct;103(4):855-9. doi: 10.1097/00000542-200510000-00025. PMID 16192779